CLINICAL TRIAL: NCT06551883
Title: Comparison of Comfort and Tolerability Between Split-dose and Single-dose Bowel Preparation Regimens Using Polyethylene Glycol Electrolyte: A Quasi-experimental Study
Brief Title: Comparison of Split-dose and Single-dose Bowel Preparation Regimens Using Polyethylene Glycol Electrolyte(PEG)
Acronym: PEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xia Wang, nurse-in-charge, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ashley
Record Dates: First submitted 2023-08-01; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bowel Preparation
Keywords: bowel preparation; compound polyethylene glycol electrolyte powder; bowel preparation quality; comfort; tolerability

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Patients in group A were given the 3L PEG in two doses: 1L of PEG was taken from 8:00 pm to 9:00 pm on the night before the examination, and the remaining 2L of PEG were taken from 4:00 am to 6:00 am on the day of the examination, with 250 mL taken every 15 minutes until finished.
  Interventions: Procedure: traditional bowel preparation regime
- Group B (Experimental): Patients in group B were given 3L of PEG in a single dose, which was taken gradually from around 3-4 am, 4-6 hours before the examination. Patients in group B were also instructed to take 250 mL every 15 minutes until the 3L were finished.
  Interventions: Procedure: different bowel preparation regime

INTERVENTIONS:
Procedure: different bowel preparation regime — Patients in Group B receive the 3L of PEG in a single dose
  Arms: Group B
Procedure: traditional bowel preparation regime — Patients in Group A receive the 3L of PEG in a split dose
  Arms: Group A

SUMMARY:
The goal of this quasi-experimental study was to compare the effect of single-dose and split-dose 3L compound polyethylene glycol electrolyte powder (PEG) regimen on the quality, comfort and tolerability of bowel preparation in patients who would undergo colonoscopy examination or treatment.

Participants in group A received a split-dose 3L PEG regimen, with 1L PEG taken on the night before the colonoscopy and 2L PEG taken 4-6 hours before the procedure. Participants in group B received a single-dose 3L PEG taken 4-6 hours before the colonoscopy.

DETAILED DESCRIPTION:
Related guidelines recommend a split-dose method for bowel preparation. However, this regimen also has limitations, such as affect patients' sleep and that of other patients in the ward, and exacerbate their discomfort due to increased hunger. This quasi-experimental study aims to investigate the effect of single-dose and split-dose 3L compound polyethylene glycol electrolyte powder (PEG) regimen on the quality, comfort and tolerability of bowel preparation.

A total of 101 patients scheduled for colonoscopy in two gastroenterology wards in a Chinese university hospital from January to June 2021 were enrolled in the study.

Patients in one department (group A) were given the 3L PEG in two doses: 1L of PEG was taken from 8:00 pm to 9:00 pm on the night before the examination, and the remaining 2L of PEG were taken from 4:00 am to 6:00 am on the day of the examination, with 250 mL taken every 15 minutes until finished. Patients in the other department (group B) were given 3L of PEG in a single dose, which was taken gradually from around 3-4 am, 4-6 hours before the examination. Patients in group B were also instructed to take 250 mL every 15 minutes until the 3L were finished.

The bowel preparation quality, comfort, sleep quality, adverse reactions, acceptance, and compliance were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* inpatients aged 18 to 70 years, with informed consent and willingness to cooperate

Exclusion Criteria:

* intestinal obstruction and stenosis;
* a history of PEG allergy;
* constipation or taking laxatives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality | The BBPS scores were filled out by the treating physician in the designated area on the patient's examination request form and were collected and organized by the research team immediately after the end of the day's clinic
  Bowel preparation quality was evaluated by the Boston Bowel Preparation Scale (BBPS)
comfort | Patients self-evaluated their comfort level during the bowel preparation process after it was completed
  a self-designed comfort evaluation scale was used, with a linear visual analog rating scale ranging from 0 (comfortable) to 4 (extremely uncomfortable).
tolerability | Patients finished the tolerability evaluation by themselves after completing bowel preparation and before being sent to the endoscopy center
  ①Patients self-assessed whether they were willing to undergo the same bowel preparation method again after the end of bowel preparation; ②Patients self-evaluated the difficulty of completing the bowel cleansing process after bowel preparation, with a score of very difficult (1 point), difficult (2 points), moderate (3 points), easy (4 points), and very easy (5 points)

SECONDARY OUTCOMES:
sleep quality | Patients finished the sleep quality evaluation by themselves after completing bowel preparation and before being sent to the endoscopy center
  Patients self-evaluated the quality of sleep on the night before bowel preparation, which is compared with usual and may be the same or slightly worse.
adherence | Patients finished the adherence evaluation by themselves after completing bowel preparation and before being sent to the endoscopy center
  Patients' compliance with medication was evaluated based on three indicators: whether the patient started taking the medication at the correct time, whether the medication was taken completely according to the instructions, and whether the patient engaged in active exercise after taking the medication

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Xia, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No